CLINICAL TRIAL: NCT01824043
Title: Pilot Study Investigating the Use of Intravitreal Ranibizumab in the Treatment of Vitreous Hemorrhage in Proliferative Diabetic Retinopathy
Brief Title: Use of Intravitreal Ranibizumab in the Treatment of Vitreous Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Regional de São José - Dr. Homero de Miranda Gomes (Other)
Responsible Party: Principal Investigator, Marcelo Brillinger Novello, Chief, Hospital Regional de São José - Dr. Homero de Miranda Gomes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUBRAHV
Record Dates: First submitted 2013-03-18; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: diabetic retinopathy; vitreous hemorrhage; intravitreal ranibizumab
MeSH Terms: conditions — Diabetic Retinopathy; Vitreous Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- vitreous hemorrhage group (Experimental): Patients will be treated monthly: intravitreal ranibizumab (0.5 mg) will be administered in an open-label fashion, using 3 monthly injections (at day 0, day 30 and day 60) followed by an additional post treatment visit, a month after the last injection, for posterior reports
  Interventions: Drug: intravitreal ranibizumab injections

INTERVENTIONS:
Drug: intravitreal ranibizumab injections — Patients will be treated monthly: intravitreal ranibizumab (0.5 mg) will be administered in an open-label fashion, using 3 monthly injections (at day 0, day 30 and day 60) followed by an additional post treatment visit, a month after the last injection, for posterior reports

SUMMARY:
Primary Objective:

To investigate the effectiveness of intravitreal applications of 0.5 mg Lucentis (ranibizumab) in patients with vitreous hemorrhage due to proliferative diabetic retinopathy.

The primary endpoint for the study will be the mean change in best-corrected visual acuity (BCVA) from baseline to the mean level at Month 3.

Secondary Objectives:

1. To assess any differences in mean change in BCVA over time;
2. To assess differences in vitreous transparency (amount of hemorrhage) with fundus angiography exam;
3. To assess any differences in retinopathy severity level according to the Early Treatment Diabetic Retinopathy Study;
4. To correlate the visual outcomes with serum glucose levels.

DETAILED DESCRIPTION:
Written informed consent must be obtained before any study assessment is performed.

This study will have only one group of patients, with a total of twenty subjects stratified based on decreased visual acuity due to vitreous hemorrhage in proliferative diabetic retinopathy:

Stratus 1 (ten subjects): patients with low to moderate diabetic vitreous hemorrhage; Stratus 2 (ten subjects): patients with severe diabetic vitreous hemorrhage. Patients will be treated monthly: intravitreal ranibizumab (0.5 mg) will be administered in an open-label fashion, using 3 monthly injections (at day 0, day 30 and day 60) followed by an additional post treatment visit, a month after the last injection, for posterior reports.

During regular, monthly visits, a detailed ophthalmologic evaluation will be performed, including a BCVA assessment. Vitreous hemorrhage density will also be assessed, according to the fundus visualization in retinal angiography:

1. low to moderate vitreous hemorrhage: posterior pole detail slightly hazy or very hazy;
2. severe vitreous hemorrhage: fundus details not visible. All patients with severe vitreous hemorrhage will have A/B ultrasound scan performed in the day of the injection. The intravitreal injection will always be the last procedure performed in a given day.

Blood samples will also be collected in each study visit, in order to assess serum glucose levels.

Laser treatment may be administered at investigator's discretion if vitreous hemorrhage reduce or disappear after the intravitreal treatment with ranibizumab to such a retinal fundus visibility level that permits photocoagulation.

All the patients of the study will be monitored about adverse events and will remain in their usual clinical and ophthalmological care after the end of the study.

Visit Schedule

Day0 Day30 Day 60 Day 90 Informed Consent X Ophthalmologic Examination X X X X Best Corrected Visual Acuity X X X X Fluorescein Angiography X X X X Serum Glucose Level X X X X A/B Ultrasound Scan X* X* X* Ranibizumab Injection X X X Laser Treatment

* ** ** ** Adverse Events Monitoring X X X X

  * Only for patients that present severe vitreous hemorrhages.
* At investigator's discretion. Check the Methodology section for details.

Population:

Patients with proliferative diabetic retinopathy with vitreous hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age who have signed an informed consent
* Patients with Type 1 or Type 2 diabetes mellitus (according to ADA or WHO guidelines).
* Patients with visual impairment due to vitreous hemorrhage.
* Medication for the management of diabetes must have been stable within 3 months prior to randomization and is expected to remain stable during the course of the study.

Exclusion criteria:

Ocular concomitant conditions/ diseases

* Concomitant conditions in the study eye which could, in the opinion of the investigator, prevent the improvement of visual acuity on study treatment
* Active intraocular inflammation (grade trace or above) in either eye
* Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye
* History of uveitis in either eye
* Ocular disorders in the study eye that may confound interpretation of study results, compromise visual acuity or require medical or surgical intervention during the 12-month study period, including retinal vascular occlusion, retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., age-related macular degeneration, ocular histoplasmosis, or pathologic myopia)
* Uncontrolled glaucoma in the study eye (according to investigator's judgment)
* Neovascularization of the iris in study eye
* Evidence of vitreomacular traction in study eye

Ocular treatments

* Panretinal laser photocoagulation in the study eye within 6 months or focal/grid laser photocoagulation in the study eye within 3 months prior to study entry
* Treatment with anti-angiogenic drugs (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc.) or intravitreal corticosteroids in either eye within 4 months prior to randomization
* Any intraocular surgery in the study eye within 3 months prior to randomization
* History of vitrectomy in study eye
* Phakic study eye with a history of intravitreal corticosteroid treatment
* Ocular conditions in the study eye that require chronic concomitant therapy with topical ocular or systemically administered corticosteroids

Systemic conditions or treatments

* History of disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, might affect the interpretation of the results of the study, or renders the patient at high risk from treatment complications
* Renal failure requiring dialysis or renal transplant OR renal insufficiency with creatinine levels >2.0 mg/dl
* Untreated diabetes mellitus
* Severe (blood pressure systolic > 160 mmHg OR diastolic > 100 mmHg) AND untreated hypertension
* Current use of or likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including Deferoxamine, Chloroquine/ hydroxychloroquine (Plaquenil), Tamoxifen, Phenothiazines and Ethambutol
* Known hypersensitivity to ranibizumab or any component of the ranibizumab formulation or to fluorescein contrast.

Compliance/ Administrative

* Previous participation in any clinical studies of investigational drugs (excluding vitamins and minerals) within 1 month (or a period corresponding to 5 half-lives of the investigational drug, whatever is longer) prior to randomization
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
* Pregnant or nursing (lactating) women.
* Inability to comply with study or follow-up procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Gain in visual acuity and transparence of vitreous in treated eyes. | 90 days

OTHER OUTCOMES:
Visual acuity improvement measured by Snellen chart | 90 days
Reduction in the ETDRS diabetic retinopathy severity level | 90 days
Serum glucose levels will be compared with the visual outcomes | 90 days
  It is expected that low glucose levels helps in better visual outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Novello, Principal Investigator — Hospital Regional Sao Jose
Locations (1):
- Marcelo Novello, São José, Santa Catarina, Brazil